CLINICAL TRIAL: NCT06902051
Title: A Prospective Study on the Application of Lateral Decubitus Position in Patients With Left Breast Cancer Undergoing Adjuvant Radiotherapy
Brief Title: Study on the Use of Lateral Decubitus Position in Left Breast Cancer Patients Undergoing Adjuvant Radiotherapy
Acronym: LDPLBC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2024-663
Record Dates: First submitted 2025-02-11; First posted 2025-03-30 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Breast Cancer; Radiotherapy; Heart protection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral Decubitus Position in Patients with Left Breast Ca (Experimental)
  Interventions: Device: Lateral Decubitus position; Device: Lateral Decubitus device
- Prone (No Intervention)

INTERVENTIONS:
Device: Lateral Decubitus position — Lateral Decubitus position with a special device
  Arms: Lateral Decubitus Position in Patients with Left Breast Ca
Device: Lateral Decubitus device — Lateral Decubitus postion with a special device
  Arms: Lateral Decubitus Position in Patients with Left Breast Ca

SUMMARY:
A Prospective Study on the Application of Lateral Decubitus Position in Patients with Left Breast Cancer Undergoing Adjuvant Radiotherapy

DETAILED DESCRIPTION:
This clinical study is a randomized, non-blind, single-center prospective clinical trial. It recruits patients with left breast cancer who are undergoing postoperative adjuvant radiotherapy. After signing the informed consent form, the clinical physician evaluates the patient's deep inspiration breath-hold (DIBH) ability and cooperation. Patients who meet the DIBH technical requirements will be randomly assigned to the DIBH supine radiotherapy group or the DIBH lateral decubitus radiotherapy group. Patients who do not meet the DIBH technical requirements will be randomly assigned to the free breathing (FB) supine radiotherapy group or the FB lateral decubitus position radiotherapy group. A total of 86 patients will be recruited. Patients who undergo lateral decubitus radiotherapy will undergo two positional fixation sessions, one in the lateral decubitus position and another one in the supine position. A CT scan will be performed in both positions. Patients using DIBH undergo scans in both FB and DIBH positions. The radiation oncologist will delineate the target area and organs at risk on the CT images, while the physicist will develop the intensity-modulated radiotherapy (IMRT) plan. After evaluating the two treatment plans, the best plan will be selected for treatment. Baseline evaluations will be completed before the radiotherapy, and follow-up evaluations will be conducted on the day of treatment completion, as well as at 3, 6, 12, 18, and 24 months after treatment. This study aims to explore the cardiac dose advantages of lateral decubitus radiotherapy in left breast cancer patients undergoing postoperative adjuvant radiotherapy. It also seeks to identify potential indicators for predicting early cardiac damage in breast cancer patients undergoing adjuvant radiotherapy. The study will effectively integrate multimodal, multidimensional feature information and multi-class models, designing a feedback mechanism to explore the risk factors associated with radiation-induced heart disease (RIHD) and predict the occurrence risk of RIHD in breast cancer patients receiving radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of the informed consent form
* Female patients aged 18-70 years
* Newly diagnosed left-sided breast cancer confirmed by histopathology
* No evidence of distant metastasis
* Undergoing modified radical mastectomy or breast-conserving surgery
* ECOG performance status of 0, 1, or 2
* Tolerance to radiotherapy
* Radiation field covering the entire left breast/chest wall ± regional lymphatic drainage area

Exclusion Criteria:

* Bilateral breast cancer at diagnosis
* History of breast reconstruction or implant placement on the affected side
* Prior radiotherapy to the chest or supraclavicular region
* Patients deemed unsuitable for the study based on the investigator's judgment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Radiotherapy Planning Dose-Volume Parameter -Volume of 5Gy heart dose | From study participation to the completion of the radiotherapy plan up to 2 years
  Volume of 5Gy heart dose
Radiotherapy Planning Dose-Volume Parameter -Max dose of LAD | From study participation to the completion of the radiotherapy plan up to 2 years
  Max dose of LAD
Radiotherapy Planning Dose-Volume Parameter -mean heart dose | From study participation to the completion of the radiotherapy plan up to 2 years
  mean heart dose
Major Cardiovascular Events | From the initiation of radiotherapy to 2 years after its completion.
  Major cardiovascular events include death due to coronary artery disease or other cardiac diseases, myocardial infarction, coronary revascularization, or hospitalization due to a major cardiovascular event (such as heart failure, valvular disease, arrhythmia, unstable angina, or other significant cardiovascular conditions).
Subclinical Cardiovascular Events- Left ventricular ejection fraction (LVEF) | From the initiation of radiotherapy to 2 years after its completion.
  Subclinical cardiovascular events include electrocardiographic abnormalities and echocardiographic abnormalities, such as:
  - Left ventricular ejection fraction (LVEF) < 50% or a reduction of > 10%.
Subclinical Cardiovascular Events- Left ventricular diastolic dysfunction | From the initiation of radiotherapy to 2 years after its completion.
  Subclinical cardiovascular events include electrocardiographic abnormalities and echocardiographic abnormalities, such as:
  - Left ventricular diastolic dysfunction, meeting at least two of the following four criteria:
  1. Mean E/e' > 14 (E/e'-lateral wall > 13 or E/Em-septum > 15).
  2. e'-lateral wall < 10 or e'-septum < 7.
  3. Tricuspid regurgitation velocity > 2.8 m/s.
  4. Left atrial volume index > 34 mL/m².

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong Provinse, China

IPD SHARING:
Plan to Share IPD: Undecided